CLINICAL TRIAL: NCT00249119
Title: Risperidone in the Treatment of Chronic Schizophrenic Patients: an International Multicentre Double-blind Parallel-group Comparative Study Versus Haloperidol.
Brief Title: A Study of the Effectiveness and Safety of Risperidone Compared With Haloperidol in Patients With Chronic Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006043
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Schizophrenia; Psychotic Disorder
Keywords: chronic schizophrenia; psychotic disorders; risperidone; antipsychotic agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of different doses of risperidone (an antipsychotic medication) compared with a fixed 10-mg dose of a standard antipsychotic, haloperidol, in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
Chronic schizophrenia is a longer-term condition that is characterized by a lack of drive, underactivity and slowness, and social withdrawal. As with the acute form of schizophrenia, delusions and hallucinations are common. This is a randomized, double-blind, parallel-group study to evaluate the effectiveness and safety of five dosages of risperidone (1, 4, 8, 12, or 16 mg per day) compared with a fixed dose of a standard antipsychotic, haloperidol (10 mg per day) in patients with chronic schizophrenia. The study is composed of two phases: a 1-week period, in which patients receive placebo and all current medication for schizophrenia treatment is stopped, and a double-blind treatment phase. The doses of study drug are increased progressively during the first week of the double blind period and then remain constant for the next 7 weeks. The primary measures of effectiveness are the percent of patients showing clinical improvement on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) and the average total PANSS score, from baseline to the end of double-blind treatment. The PANSS is a rating scale that measures the symptoms of schizophrenia. Safety evaluations include the incidence of adverse events, results of clinical laboratory tests (hematology, biochemistry, urinalysis, and hormone levels), plasma levels of risperidone, measurements of vital signs and body weight, physical examination and electrocardiogram (ECG) findings, neurological examinations, and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone doses of 4, 8, 12, or 16 mg/day are more effective than risperidone 10 mg/day, as measured by clinical improvement on PANSS and the average total score for PANSS, in patients with chronic schizophrenia. Risperidone oral tablets, twice-daily, starting with 1 or 2 mg/day, increasing gradually in Week 1 (except for 1 mg/day group), then 0.5, 2, 4, 6, or 8 mg twice daily for 7 weeks. Haloperidol oral tablets, twice-daily, starting with 2 mg/day, increasing to 5 mg twice daily in Week 1, then 5 mg twice daily for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic schizophrenic disorder, according to the Diagnostic and Statistical Manual of Mental Diseases, 3rd edition (DSM-III-R) criteria
* total score on the PANSS at study entry of >=60 and <=120
* physical and neurological examination and ECG findings and clinical hematology, biochemistry, and urinalysis test results within normal limits before study entry
* patients must be able to be hospitalized the first 3 weeks of the study, if possible.

Exclusion Criteria:

* Patients with mental disorders other than chronic schizophrenic disorder
* patients with clinically significant organic or neurologic diseases
* women who are pregnant or breastfeeding, and women of childbearing potential without adequate birth control measures
* patients with epilepsy
* history of alcohol or drug abuse history within the previous 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1579 (Actual)
Dates: Study Completion 1991-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients showing clinical improvement, defined as a >=20% reduction in the total PANSS score from baseline to end of double-blind treatment, and the mean change from baseline to end of double-blind treatment in total PANSS score.

SECONDARY OUTCOMES:
Mean PANSS Positive Subscale Score; Mean PANSS Negative Subscale Score; mean PANSS General Psychopathology Subscale Score; mean separate PANSS item scores; safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Result] Peuskens J. Risperidone in the treatment of patients with chronic schizophrenia: a multi-national, multi-centre, double-blind, parallel-group study versus haloperidol. Risperidone Study Group. Br J Psychiatry. 1995 Jun;166(6):712-26; discussion 727-33. doi: 10.1192/bjp.166.6.712. PMID 7545060